CLINICAL TRIAL: NCT05777603
Title: Phase I Study of Aerosolized Antibiotics and Pembrolizumab in Advanced Non-Small Cell Lung Cancer
Brief Title: Study of Aerosolized Antibiotics and Pembrolizumab in Advanced Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10001516; 001516-C
Record Dates: First submitted 2023-03-18; First posted 2023-03-21 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01-08

CONDITIONS: Advanced Non Small Cell Lung Cancer
Keywords: Immune Checkpoint Inhibitor; lung microbiota; anti-PD1 antibody; inhaled antibiotic
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Pembrolizumab + de-escalating doses of aztreonam and vancomycin
  Interventions: Drug: aerosolized aztreonam; Drug: aerosolized vancomycin; Drug: pembrolizumab

INTERVENTIONS:
Drug: aerosolized aztreonam — antibiotic with gram-negative bacteria coverage
Drug: aerosolized vancomycin — antibiotic with gram-positive bacteria coverage
Drug: pembrolizumab — standard of care therapy/monoclonal antibody for patients with advanced NSCLC

SUMMARY:
Background:

Non-small cell lung cancer (NSCLC) can be hard to treat and is often fatal. People with NSCLC commonly have changes in the bacteria that populate their lungs. These bacterial changes may aid tumor growth. Researchers want to find out if treating the bacteria, too, can help cancer treatment work better.

Objective:

To test 2 inhaled antibiotics (aztreonam and vancomycin), combined with a standard cancer treatment, in people with NSCLC.

Eligibility:

People aged 18 years and older with NSCLC that has returned or progressed after treatment and cannot be treated with surgery.

Design:

Participants will be screened. They will have a physical exam with blood tests. They may blow into a machine to test how well their lungs work. They will have imaging scans. They may need to have a small piece of tissue cut from their tumor (biopsy).

Participants will be treated in six 21-day cycles. They will visit the clinic to receive a drug for cancer treatment on the first day of each cycle. This drug will be administered through a tube attached to a needle inserted into a vein in the arm.

The 2 antibiotic drugs will be in the form of a fine mist that can be inhaled. Participants use a device to take these drugs at home. They will inhale aztreonam up to 3 times a day and vancomycin 1 or 2 times a day. They will take these drugs during only 3 of the treatment cycles.

Biopsies and other tests will be repeated halfway through and after the study treatment.

Follow-up visits will continue for 1 year after study treatment.

DETAILED DESCRIPTION:
Background:

* Dysbiosis of the lung microbiome is commonly seen in patients with advanced non-small cell lung cancer (NSCLC). It is associated with increased bacterial burden and decreased bacterial diversity in tumors
* Preclinical studies using genetically engineered mouse (GEM) models show that dysbiosis of the lung microbiome promotes tumor growth in NSCLC

Objective:

- To assess the safety of combined aerosolized antibiotics (aztreonam and vancomycin) with pembrolizumab IV, in participants with advanced NSCLC

Eligibility:

* Histological confirmation of NSCLC that is not amenable to surgery
* Disease has progressed after FDA-approved frontline therapy for NSCLC
* PD-L1Tumor Proportion Score (TPS) >=1% detected at any time since diagnosis.
* Measurable and progressive disease
* Age >=18 years
* ECOG performance status <=2
* Participants must have adequate organ and bone marrow function

Design:

* This is a phase I, open-label, single-arm study evaluating the safety and feasibility of combined aerosolized antibiotics (aztreonam and vancomycin) and pembrolizumab in advanced NSCLC
* Participants will be given six cycles of treatments; each cycle is three weeks (21 days)
* Participants receive pembrolizumab 200mg IV on Day 1 of each cycle
* During cycles 1, 3 and 5, participants will self-administer aerosolized aztreonam 3 times a day and vancomycin twice a day from Day 2 through Day 21
* There are two dose levels of aerosolized antibiotics: participants start with Dose Level 1 (aztreonam 75mg three times a day and vancomycin 250mg twice a day)
* If participants cannot tolerate Dose Level 1, treatment will be de-escalated to Dose Level
* 1 (aztreonam 75mg once a day and vancomycin 250mg once a day)
* Participants will be enrolled based on "3+3" scheme to test the primary endpoints of safety and feasibility
* Up to 18 evaluable participants will be enrolled

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Histologically or cytologically non-small cell lung cancer confirmed by outside pathology report or via the Laboratory of Pathology, NCI.
2. Have measurable disease, per RECIST 1.1, that is not amenable to surgery.
3. PD-L1 Tumor Proportion Score (TPS) >=1% detected at any time since diagnosis, based on a pathology report from an outside hospital or Laboratory of Pathology, NCI. PD- L1 expression testing must be conducted using one of the FDA approved diagnostic devices listed here: https://www.fda.gov/medical-devices/in-vitro-diagnostics/list- cleared-or-approved-companion-diagnostic-devices-in-vitro-and-imaging-tools.
4. Patient s disease has progressed after FDA-approved frontline therapy for NSCLC.
5. Age >=18 years.
6. ECOG performance status <=2.
7. Must have adequate organ and marrow function as defined below:

   * Leukocytes >=3,000/mcL
   * absolute neutrophil count >=1,500/mcL
   * platelets >=100,000/mcL
   * total bilirubin<TAB>within normal institutional limits
   * AST/ALT <=2.5 X institutional upper limit of normal
   * creatinine clearance >=60 mL/min/1.73 m^2 (calculated based on CKD-EPI formula or directly measured) for participants with creatinine levels above institutional normal.
8. Participants with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression.
9. Participants with new or progressive brain metastases (active brain metastases) are eligible if immediate CNS specific treatment is not required per standard of care and is unlikely to be required during the first cycle of therapy.
10. Human immunodeficiency virus (HIV)-infected participants on effective anti-retroviral therapy with undetectable viral load within the 6 months before study treatment initiation are eligible for this trial.
11. For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
12. Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
13. Individuals of child-bearing potential (IOCBP) must agree to use effective contraception (e.g., hormonal intrauterine device [IUD], tubal ligation, partner has had prior vasectomy) beginning at study entry until 4 months after the completion of therapy. Note: abstinence, defined as no heterosexual sexual intercourse when this is in line with the preferred and usual lifestyle of the participant, is also acceptable.
14. Breastfeeding participants must be willing to discontinue breastfeeding for the duration of study treatment.
15. Ability of participant to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

1. Participants who are receiving any other investigational agents.
2. Participants with ongoing Epstein-Barr virus or cytomegalovirus infection
3. History of allergic reactions attributed to compounds of similar chemical or biologic composition to pembrolizumab, aztreonam, vancomycin and albuterol.
4. Pregnancy (confirmed with beta-HCG serum or urine pregnancy test performed in individuals of childbearing potential at screening).
5. Pulmonary function FEV1 (Forced Expiratory Volume in the first second) <25% will be excluded based on the requirement of receiving aerosolized aztreonam.
6. History of severe immune-related adverse events (irAEs), defined as any grade neurological or cardiac irAEs, any grade 3 or 4 irAE (except fully controlled endocrine irAEs with appropriate hormone supplementation), and any grade pneumonitis.
7. Uncontrolled intercurrent illness that would limit compliance with study requirements.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLTs) - type and grade | Start of therapy through 1 year after last study drug dose
  Safety will be evaluated by reported grades of toxicities, including DLTs at each dose levels.

SECONDARY OUTCOMES:
Dose limiting toxicities (DLTs) - type and grade | Start of therapy through 1 year after last study drug dose.
  Recommended phase 2 dose will be determined by reported grades of toxicities, including DLTs at each dose levels.
Fraction of participants who received adequate doses of all agents at each dose level | Between start of therapy through 1 year after last study drug dose.
  Feasibility will be reported as the fraction of participants who receive adequate doses of all drug agents without DLT at each dose level.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Zhao, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
-- All IPD recorded in the medical record will be shared with intramural investigators upon request. -- All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: -- Clinical data available during the study and indefinitely. -- Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: -- Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. -- Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001516-C.html